CLINICAL TRIAL: NCT00610402
Title: Incidence of Ocular Antibodies in Patients With Sturge - Weber Syndrome (SWS)
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Mainz University (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Other Study IDs: 20065691
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Sturge - Weber Syndrome (SWS)
MeSH Terms: conditions — Brain Stem Infarctions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample tear drop sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- blood sample tear drop sample: blood sample tear drop sample
  Interventions: Other: blood sample tear drop sample

INTERVENTIONS:
Other: blood sample tear drop sample — blood sample tear drop sample

SUMMARY:
Sturge-Weber Syndrome (SWS) is a neurological disorder characterized at birth by seizures and a large port-wine stain birthmark on the forehead and upper eyelid of one side of the face. SWS is also accompanied by an increased pressure within the eye (glaucoma) which can develop very early in life.

Glaucoma represents a group of ocular disorders that are characterized by the loss of retinal ganglion cells and their axons, damage to the optic nerve, and gradual loss of visual field. Recently, several studies provided evidence that there is a potential role of the immune system in the pathogenesis of glaucoma.

These findings suggest that there might be changes in systemic humoral immunity possibly underlying the optic neuropathy in at least some glaucoma patients.

DETAILED DESCRIPTION:
The ocular antibody profile in patients with SWS is unknown.The researchers want to study on blood and tear drop samples from patients with SWS to determine the incidence of ocular antibodies in patients with this syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers with SWS of all ages

Exclusion Criteria:

* Volunteers without SWS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2007-07; Primary Completion 2007-07 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D,PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States